CLINICAL TRIAL: NCT02302638
Title: Embryo Development and Utilization Using Two Commercial Single-step Media
Brief Title: Embryo Development Using Two Commercial Single-step Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sage vs CSCM
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: single-step media; embryo development; blastocyst formation; embryo utilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sage 1-step (Active Comparator): Embryo culture in different single-step media:
  Half of each patient's oocytes will be randomly allocated to be cultured in Sage 1-step medium for up to six days following oocyte retrieval.
  Interventions: Other: embryo culture in different single-step media
- CSCM (Active Comparator): Embryo culture in different single-step media:
  Half of each patient's oocytes will be randomly allocated to be cultured in CSC medium for up to six days following oocyte retrieval.
  Interventions: Other: embryo culture in different single-step media

INTERVENTIONS:
Other: embryo culture in different single-step media — Half of each patient's oocytes will be randomly allocated to be cultured either in Sage 1-step medium (Origio) or in CSC medium (Irvine Scientific) for up to six days following oocyte retrieval.

SUMMARY:
This prospective study with sibling oocytes will evaluate the efficiency of two commercial single-step media, namely Sage 1-step and Continuous Single Culture Medium (CSCM), in terms of embryo utilization rates, blastocyst formation rates, embryo quality and pregnancy rates. Embryos will be cultured continuously for up to 6 days under identical conditions.

ELIGIBILITY:
Inclusion Criteria:

* at least 10 oocytes retrieved

Exclusion Criteria:

* frozen oocytes
* testicular biopsy
* less than 10 oocytes retrieved
* older than 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Utilization rates | 6 days post oocyte retrieval
  Utilization = embryos selected for transfer and cryopreservation
Blastocyst formation | 5 days post oocyte retrieval
  Number of blastocysts on day 5 post oocyte retrieval per fertilized oocytes

SECONDARY OUTCOMES:
Embryo quality on day 3 | 3 days post oocyte retrieval
blastocyst quality on day 5 | 5 days post oocyte retrieval
positive pregnancy test | 15 days post oocyte retrieval
clinical pregnancy | 7 weeks of gestation
  presence of gestational sac with positive fetal heartbeat

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis A Sfontouris, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia Assisted Reproduction Unit, Athens, Attica, Greece

REFERENCES:
- [Derived] Sfontouris IA, Kolibianakis EM, Lainas GT, Venetis CA, Petsas GK, Tarlatzis BC, Lainas TG. Blastocyst utilization rates after continuous culture in two commercial single-step media: a prospective randomized study with sibling oocytes. J Assist Reprod Genet. 2017 Oct;34(10):1377-1383. doi: 10.1007/s10815-017-0997-0. Epub 2017 Jul 17. PMID 28718081